CLINICAL TRIAL: NCT02546284
Title: A Phase 1 Study of Lenzilumab in Subjects With Previously Treated Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Study of Lenzilumab in Previously Treated Patients With Chronic Myelomonocytic Leukemia (CMML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGEN003-05
Record Dates: First submitted 2015-08-27; First posted 2015-09-10 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Chronic Myelomonocytic Leukemia (CMML)
Keywords: CMML
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — lenzilumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Agent lenzilumab (Experimental): Dose levels: lenzilumab IV infusion once monthly for a 28 day dosing cycle (with extra dose on Day 15 during cycle). Three (3) to Six (6) subjects will be enrolled into planned escalating cohorts of 200 mg, 400 mg or 600 mg lenzilumab.
  Interventions: Drug: lenzilumab

INTERVENTIONS:
Drug: lenzilumab
  Other Names: Monoclonal Antibody

SUMMARY:
This is a multicenter, open-label, repeat-dose, Phase 1 Dose Escalation Study to evaluate safety, pharmacokinetics, and clinical activity.

DETAILED DESCRIPTION:
The purpose of the study is to examine the safety and determine the recommended Phase 2 dose of lenzilumab when administered to subjects with previously treated CMML who meet the entry criteria. Study will begin enrollment in July 2016.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CMML
* CMML that is refractory to, or progressed following treatment with a hypomethylating agent or other standard of care treatment
* Eastern Cooperative Oncology Group (ECOG) score ≤ 2
* Able to provide bone marrow biopsy samples
* Acceptable laboratory results

Exclusion Criteria:

* Leukemia other than CMML
* Recent chemotherapy or radiation therapy (within 14 days before first dose of lenzilumab)
* Concurrent use of human granulocyte-macrophage colony-stimulating factor
* Pregnant or breastfeeding
* Know HIV virus infection
* History of another malignancy within the past 2 years (some skin cancer and prostate cancers permitted)
* Significant intercurrent illness
* History or current diagnosis of Pulmonary Alveolar Proteinosis or Hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Safety of lenzilumab (as measured by the number of participants with adverse events) at various doses in order to determine a recommended Phase 2 dose | Up to an average of 12 months

SECONDARY OUTCOMES:
Clinical activity of lenzilumab (as measured by changes in spleen size, blood and bone marrow measurements of disease, clinical symptoms, etc) | Up to an average of 12 months

OTHER OUTCOMES:
Maximum plasma concentration (Cmax) of lenzilumab | At end of infusion or 1 hour after end of infusion on Day 1
Time to maximum plasma concentration (Tmax) of lenzilumab | Pre-dose to end of infusion or 1 hour after end of infusion on Day 1
Minimum plasma concentration (Cmin) of lenzilumab | At Day 15
Area under the plasma concentration curve (AUC) of lenzilumab | Predose, end of infusion, 1 hour after end of infusion on Day 1, Day 2, Day 7, Day 15
Plasma half life (t ½) of lenzilumab | End of infusion, 1 hour after end of infusion on Day 1, Day 2, Day 7, Day 15
Plasma clearance (CL) of lenzilumab | End of infusion, 1 hour after end of infusion on Day 1, Day 2, Day 7, Day 15
lenzilumab immunogenicity (as measured by antibodies against lenzilumab in blood) | Up to an average of 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic Cancer Center Clinical Research, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No